CLINICAL TRIAL: NCT01928433
Title: A Multi-Dose, Double-Blind, Double-Dummy, Active- Control, Randomized Clinical (Phase II) Study of Two Dosing Regimens of Finafloxacin for the Treatment of cUTI and/or Acute Pyelonephritis Requiring Hospitalisation.
Brief Title: Finafloxacin for the Treatment of cUTI and/or Acute Pyelonephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MerLion Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FINA-007; 2011-006041-14 (EudraCT Number)
Record Dates: First submitted 2013-07-17; First posted 2013-08-26 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Urinary Tract Infections; Acute Pyelonephritis
Keywords: Urinary Tract Infection; Pyelonephritis
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis | interventions — finafloxacin; Sodium Chloride; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Finafloxacin 5 days (Experimental): Intervention:
  Finafloxacin 800 mg i.v. once daily and Ciprofloxacin placebo i.v. twice daily. Finafloxacin 800 mg tablets once daily and Ciprofloxacin placebo oral twice daily Finafloxacin verum (i.v. and oral) for a total of 5 days.
  Interventions: Drug: Finafloxacin 800 mg i.v. once daily; Drug: Finafloxacin 800 mg tablets once daily; Drug: Ciprofloxacin placebo i.v. twice daily; Drug: Ciprofloxacin placebo oral twice daily
- Finafloxacin 10 days (Experimental): Intervention:
  Finafloxacin 800 mg i.v. once daily and Ciprofloxacin placebo i.v. twice daily. Finafloxacin 800 mg tablets once daily and Ciprofloxacin placebo oral twice daily Finafloxacin verum (i.v. and oral) for a total of 10 days.
  Interventions: Drug: Finafloxacin 800 mg i.v. once daily; Drug: Finafloxacin 800 mg tablets once daily; Drug: Ciprofloxacin placebo i.v. twice daily; Drug: Ciprofloxacin placebo oral twice daily
- Ciprofloxacin 10 days (Active Comparator): Intervention:
  Ciprofloxacin 400 mg i.v. twice daily and Finafloxacin placebo i.v. once daily Ciprofloxacin 500 mg oral twice daily and Finafloxacin placebo tablets once daily Ciprofloxacin (i.v. and oral) for a total of 10 days.
  Interventions: Drug: Finafloxacin placebo i.v. once daily; Drug: Finafloxacin placebo tablets once daily; Drug: Ciprofloxacin 400 mg i.v. twice daily; Drug: Ciprofloxacin 500 mg oral twice daily

INTERVENTIONS:
Drug: Finafloxacin 800 mg i.v. once daily — Infused over 60 mins [i.v. pump]) for at least 3 days.
  Other Names: Finafloxacin
  Arms: Finafloxacin 10 days; Finafloxacin 5 days
Drug: Finafloxacin placebo i.v. once daily — Infused over 60 mins [i.v. pump]) for at least 3 days.
  Other Names: Saline
  Arms: Ciprofloxacin 10 days
Drug: Finafloxacin 800 mg tablets once daily — Administered as four 200 mg tablets
  Other Names: Finafloxacin
  Arms: Finafloxacin 10 days; Finafloxacin 5 days
Drug: Finafloxacin placebo tablets once daily — Administered as four tablets
  Arms: Ciprofloxacin 10 days
Drug: Ciprofloxacin 400 mg i.v. twice daily — Infused over approximately 60 mins [i.v. pump]) for at least 3 days
  Other Names: Ciprofloxacin Kabi Infusionslösung
  Arms: Ciprofloxacin 10 days
Drug: Ciprofloxacin placebo i.v. twice daily — Infused over approximately 60 mins [i.v. pump]) for at least 3 days
  Other Names: Saline
  Arms: Finafloxacin 10 days; Finafloxacin 5 days
Drug: Ciprofloxacin 500 mg oral twice daily — Administered as two 250 mg capsules.
  Other Names: Ciprofloxacin real 250/500/750 mg
  Arms: Ciprofloxacin 10 days
Drug: Ciprofloxacin placebo oral twice daily — Administered as two capsules.
  Arms: Finafloxacin 10 days; Finafloxacin 5 days

SUMMARY:
The primary objective of this study is to evaluate the microbiological and clinical outcome of treatment with finafloxacin for 5 days versus finafloxacin for 10 days versus ciprofloxacin for 10 days as a reference comparator.

Finafloxacin shows increased activity in an acidic environment which is associated with indications such as uUTI and cUTI. Given the acidic pH of urine and concentration of finafloxacin excreted via the urinary tract in humans it should be proven if the finafloxacin treatments offer significant advantages over the currently available treatments for UTI.

DETAILED DESCRIPTION:
Fluoroquinolones are frequently prescribed for complicated Urinary Tract Infections (cUTI) and pyelonephritis, due to their activity against cUTI pathogens and high levels of excretion in the urine following oral and i.v. administration. However, many currently prescribed fluoroquinolones exhibit reduced antibacterial activity at low pH, which suggests reduced activity in infected urinary tracts.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female subjects ≥ 18 years of age.
2. If a female and

   1. subject is of childbearing potential, must have documented use of using an effective contraceptive method (such as IUD, hormonal birth control, condom and spermicidal jelly, etc.) during the study, Contraception must have been used for at least 2 months before starting the study. A documented negative urine pregnancy test must be provided and the subject must be non-lactating.
   2. subject is of non-childbearing potential, must be post-menopausal (i.e. has had amenorrhea for a minimum of 12 consecutive months) or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
   3. subject is truly abstinent. This is accepted as a method of contraception, but only when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
3. If a male, should agree to use reliable birth control methods (contraception or other barrier device) during study participation.
4. Must have complicated lower urinary tract infection or acute complicated or uncomplicated pyelonephritis (cPN or uPN; see section 5.3) and must have at least two of the following acute signs and symptoms

   1. Chills or rigors or warmth associated with fever (e.g. oral temperature greater than 38.0 degrees Celsius ).
   2. Flank pain (pyelonephritis) or pelvic pain (cUTI).
   3. Nausea or vomiting.
   4. Dysuria, urinary frequency, or urinary urgency.
   5. Costo-vertebral angle tenderness (pyelonephritis) on physical examination.
5. Provide one pre-treatment adequate urine sample (the urine sample must return a positive culture in order for the subject to remain eligible for the study) For males: midstream clean catch, for females: in-out catheterisation or midstream clean catch. The urine sample must be provided within 24 hours before the start of administration of the first dose of study drug.

   A positive urine culture is defined as:
   * ≥ 105 CFU/mL of one causative pathogen in the case of cUTI
   * ≥ 104 CFU/mL of one causative pathogen in case of Pyelonephritis

   A negative urine culture is defined as:
   * < 105 CFU/mL of causative pathogen/s and/or non-target pathogens at any number of CFUs in the case of cUTI
   * < 104 CFU/mL of causative pathogen/s and/or non-target pathogens at any number of CFUs in the case of Pyelonephritis Patients may be admitted to the study pending baseline urine culture results. Treatment should NOT be delayed pending urine culture results.

   NOTE: Because biofilms on indwelling catheters (e.g. Foley catheters) are more likely to be present after the catheter has been in place for a period of time, samples should be collected following the placement of a new catheter. If the placement of a new catheter is contraindicated or is not feasible, specimens should be collected using aseptic techniques with the urine obtained through a properly disinfected collection port. Urine samples should never be obtained from the collection bag.

   If the subject's pre-treatment culture shows the presence of a ciprofloxacin resistant pathogen the Investigator has to decide according to clinical signs and symptoms whether the subject can stay in the study.

   In the event of a negative urine culture, the subject must be withdrawn from the study and switched to standard care, because the inclusion criterion is not fulfilled.

   A urine culture is defined as contaminated if:
   * at least one causative pathogen with ≥ 105 CFU/mL is present AND at least one non-pathogen or additional causative pathogen/s at any number of CFU/mL are present in the case of cUTI
   * at least one causative pathogen with ≥ 104 CFU/mL is present AND at least one non-pathogen or additional causative pathogen/s with any number of CFU/mL in the case of pyelonephritis Subjects with contaminated urine cultures will be permitted to continue in the study, although this will impact on the subject's eligibility for analysis (see section 9.3).
6. Have pyuria (i.e. a dipstick analysis positive for leukocyte esterase or at least 10 white blood cells per cubic millimetre [1 µl]).
7. Be considered ill enough to be hospitalized for at least 3 days and require initial parenteral therapy to manage cUTI and/or acute pyelonephritis by the standard of care.
8. Provide written informed consent to participate in the study.
9. Be willing and able to comply with all study procedures and activities.

Exclusion Criteria:

1. Uncomplicated cystitis in females.
2. Failed previous antibiotic treatment within the last 4 weeks due to culture confirmed fluoroquinolone resistant pathogens.
3. Having ileal loops, urinary diversion with bowel segments or suspected or confirmed vesico-ureteral reflux, suspected or confirmed perinephric or intrarenal abscess (if an abscess is suspected an ultrasound should be performed to confirm and exclude).
4. History of renal transplant any permanent complicating factors of the urinary tract (including complete obstruction, suspected or confirmed prostatitis or epididymitis) which cannot be effectively treated during the therapy of the infection.
5. Indwelling urinary catheters expected to remain in place after therapy has been completed.
6. The urinary tract infection or any other concomitant bacterial infection that requires systemic antibiotic therapy (in addition to the study treatment) at the time of randomisation. Antibiotics with only gram-positive activity are permitted.
7. Any infection that, in the opinion of the Investigator, would be considered intractable and likely to require more than 10 days of study drug therapy.
8. Any recent use (e.g., within 48 hours before the first dose of study medication) of an antimicrobial therapy with a drug that has activity in the treatment of urinary tract infection.
9. Having been exposed to any fluoroquinolone in the 30 days before Day 1 (study enrolment), previous participation in a finafloxacin clinical trial or participation within the last 30 days in any other clinical study in general.
10. In the 12 months before study enrolment: known uncontrolled condition of hypertension or symptomatic hypotension, known uncontrolled cardiac arrhythmia, known ischaemic heart disease or history of myocardial infarction, coronary artery bypass surgery or percutaneous transluminal coronary angioplasty.
11. Significantly immunocompromised (defined as a WBC < 1000) and/or having a known infection with human immunodeficiency virus (HIV/AIDS), any haematological malignancy, bone marrow transplantation, or current immunosuppressive therapy (including but not limited to cancer chemotherapy, or medications for prevention of organ transplantation rejection).
12. Any concomitant psychiatric, neurological or behavioural disorder, including epilepsy or other lesions of the central nervous system sufficient in the opinion of the Investigator to prevent or compromise the subject's participation in the study.
13. Any known concomitant bacterial or fungal sexually transmitted disease with the exception of candidiasis.
14. Having, in the opinion of the Investigator, any clinically significant serious or unstable physical illness likely to impact on the subject's wellbeing or the conduct and analysis of the study, including, but not limited to, acute hepatic failure, respiratory failure, severe, persistent diarrhoea and septic shock.
15. Any surgical or medical condition which might interfere with the distribution, metabolism or excretion of the drug, including, but not limited to moderate (including estimated creatinine clearance of 30 - 59 mL/min) or severe impairment of renal function (including an estimated creatinine clearance of < 30 mL/min), requirement for peritoneal dialysis, haemodialysis or haemofiltration, or oliguria.
16. Any malignant disease or a history of malignant neoplasm requiring a treatment with immune suppressive properties in the 6 months before baseline.
17. Known history of drug abuse.
18. Clinically abnormal haematology, biochemistry and urinalysis results at baseline including, but not limited to:

    * AST, ALT, or alkaline phosphatase level greater than 3 times the upper limit of normal (ULN).
    * Total bilirubin greater than 2 times ULN.
    * WBC count less than 1000/μL, platelet count less than 50,000/μL.
    * Haematocrit less than 25%.
    * Creatinine clearance < 60mL/minute.
19. Any clinically significant ECG abnormality on the baseline ECG subjects at risk for torsade de pointes arrhythmia or a history of significant or inadequately treated cardiac disease.
20. Documented history of hypersensitivity or allergy to or known contraindication to the use of fluoroquinolones.
21. Any history of tendon lesions or ruptures either during quinolone treatment or for any other reason.
22. Concomitant tizanidine use.
23. Any administration of corticosteroids equivalent to or greater than 20 mg of prednisone per day for more than 14 days before randomisation.
24. The subject, planned to be enrolled is an employee or relative of any involved study Investigator or any involved institution including MerLion or Galenus.
25. Life expectancy of less than 3 months.
26. Women who are pregnant or nursing.
27. Any other condition that, in the opinion of the Investigator, would prevent the subject from effectively participating in the study, place the subject at risk or affect the assessment of efficacy and safety of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Wagenlehner, Prof., Principal Investigator — Germany: University Hospital Giessen and Marburg, Department of Urology; Michal Nowicki, Prof., Principal Investigator — Poland: Medical University Lodz, Department of Nephrology
Locations (1):
- Universitätsklinikum Giessen, Klinik für Urologie, Kinderurologie und Andrologie, Giessen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wagenlehner F, Nowicki M, Bentley C, Luckermann M, Wohlert S, Fischer C, Vente A, Naber K, Dalhoff A. Explorative Randomized Phase II Clinical Study of the Efficacy and Safety of Finafloxacin versus Ciprofloxacin for Treatment of Complicated Urinary Tract Infections. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e02317-17. doi: 10.1128/AAC.02317-17. Print 2018 Apr. PMID 29339395
- [Derived] Taubert M, Luckermann M, Vente A, Dalhoff A, Fuhr U. Population Pharmacokinetics of Finafloxacin in Healthy Volunteers and Patients with Complicated Urinary Tract Infections. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e02328-17. doi: 10.1128/AAC.02328-17. Print 2018 Apr. PMID 29339394
- [Derived] Vente A, Bentley C, Luckermann M, Tambyah P, Dalhoff A. Early Clinical Assessment of the Antimicrobial Activity of Finafloxacin Compared to Ciprofloxacin in Subsets of Microbiologically Characterized Isolates. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e02325-17. doi: 10.1128/AAC.02325-17. Print 2018 Apr. PMID 29339393

RESULTS

PARTICIPANT FLOW:
Groups:
- Finafloxacin 5 Days: Finafloxacin (i.v. and oral) for a total of 5 days.
  Finafloxacin 800 mg i.v. once daily
  Finafloxacin 800 mg tablets (as four 200 mg tablets) once daily
  Ciprofloxacin placebo i.v. two times daily
  Ciprofloxacin placebo oral (as two capsules each) two times daily
- Finafloxacin 10 Days: Finafloxacin (i.v. and oral) for a total of 10 days.
  Finafloxacin 800 mg i.v. once daily
  Finafloxacin 800 mg tablets (as four 200 mg tablets) once daily
  Ciprofloxacin placebo i.v. two times daily
  Ciprofloxacin placebo oral (as two capsules each) two times daily
- Ciprofloxacin 10 Days: Ciprofloxacin (i.v. and oral) for a total of 10 days.
  Finafloxacin placebo i.v. once daily
  Finafloxacin placebo tablets (as four tablets) once daily
  Ciprofloxacin 400 mg i.v. two times daily
  Ciprofloxacin 500 mg oral (as two 250 mg capsules) two times daily
Period: Overall Study
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days
Started | 76 | 75 | 74
Completed | 56 | 54 | 46
Not Completed | 20 | 21 | 28
Not completed — Adverse Event | 5 | 2 | 5
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Lack of Efficacy | 5 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 4 | 0
Not completed — Negative screening urine culture | 7 | 6 | 10
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Other reasons | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Subjects that received at least one dose of study medication (safety set).
Groups:
- Total: Total of all reporting groups
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days | Total
Number analyzed (Participants) | 76 | 75 | 72 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 43 | 48 | 143
  >=65 years | 24 | 32 | 24 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (19.63) | 58.0 (19.28) | 51.0 (21.01) | 54.6 (20.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 62 | 57 | 183
  Male | 12 | 13 | 15 | 40
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 14 | 7 | 31
  Poland | 66 | 61 | 65 | 192

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical and Microbiological Response
Description: The primary endpoint of this study is the clinical and microbiological response of patients with cUTI or pyelonephritis to treatment with finafloxacin for 5 days versus finafloxacin for 10 days versus ciprofloxacin for 10 days as a reference comparator at the Test of Cure (ToC) visit (Day 17) in the microbiological intent-to-treat population (micro-ITT population).
  Clinical response is defined as resolution of the symptoms of cUTI present at trial entry and no new symptoms developed. Microbiological response is defined as elimination or reduction of study entry pathogens to ≤ 10e3 CFU/mL on urine culture. The clinical and microbiological response will be assessed for each group on Day 17 and will be compared between the three groups to assess the efficacy in each group.
Time Frame: Day 17
Population: The micro-ITT population is composed of all randomized patients who have a baseline bacterial pathogen on culture of urine or blood that causes UTI against which the investigational drug has antibacterial activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days
Number analyzed (Participants) | 64 | 68 | 61
Participants | 45 | 46 | 35

2. Secondary Outcome: Number of Participants With Clinical and Microbiological Response at the On Therapy (OT) Visit (Day 3).
Description: The clinical and microbiological response as the efficacy parameter will be assessed for each group and will be compared between the three groups. Separate analyses will be performed for all time points for the clinical and microbiological responders and compared also between the different groups.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Finafloxacin 5 Days: Intervention:
  Finafloxacin 800 mg i.v. once daily and Ciprofloxacin placebo i.v. twice daily. Finafloxacin 800 mg tablets once daily and Ciprofloxacin placebo oral twice daily Finafloxacin verum (i.v. and oral) for a total of 5 days.
  Finafloxacin 800 mg i.v. once daily: Infused over 60 mins [i.v. pump]) for at least 3 days.
  Finafloxacin 800 mg tablets once daily: Administered as four 200 mg tablets
  Ciprofloxacin placebo i.v. twice daily: Infused over approximately 60 mins [i.v. pump]) for at least 3 days
  Ciprofloxacin placebo oral twice daily: Administered as two capsules.
- Finafloxacin 10 Days: Intervention:
  Finafloxacin 800 mg i.v. once daily and Ciprofloxacin placebo i.v. twice daily. Finafloxacin 800 mg tablets once daily and Ciprofloxacin placebo oral twice daily Finafloxacin verum (i.v. and oral) for a total of 10 days.
  Finafloxacin 800 mg i.v. once daily: Infused over 60 mins [i.v. pump]) for at least 3 days.
  Finafloxacin 800 mg tablets once daily: Administered as four 200 mg tablets
  Ciprofloxacin placebo i.v. twice daily: Infused over approximately 60 mins [i.v. pump]) for at least 3 days
  Ciprofloxacin placebo oral twice daily: Administered as two capsules.
- Ciprofloxacin 10 Days: Intervention:
  Ciprofloxacin 400 mg i.v. twice daily and Finafloxacin placebo i.v. once daily Ciprofloxacin 500 mg oral twice daily and Finafloxacin placebo tablets once daily Ciprofloxacin (i.v. and oral) for a total of 10 days.
  Finafloxacin placebo i.v. once daily: Infused over 60 mins [i.v. pump]) for at least 3 days.
  Finafloxacin placebo tablets once daily: Administered as four tablets
  Ciprofloxacin 400 mg i.v. twice daily: Infused over approximately 60 mins [i.v. pump]) for at least 3 days
  Ciprofloxacin 500 mg oral twice daily: Administered as two 250 mg capsules.
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days
Number analyzed (Participants) | 64 | 68 | 61
Participants | 39 | 40 | 33

3. Secondary Outcome: Number of Participants With Clinical and Microbiological Response at the End of Therapy (EoT) Visit (Day 10).
Description: as for outcome 2
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days
Number analyzed (Participants) | 64 | 68 | 61
Participants | 49 | 49 | 44

4. Secondary Outcome: Number of Participants With Clinical and Microbiological Response at the End of Study (EoS) Visit (Day 24).
Description: as for outcome 2
Time Frame: Day 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days
Number analyzed (Participants) | 64 | 68 | 61
Participants | 47 | 42 | 34

5. Secondary Outcome: The Safety and Tolerability of Multiple Doses of Finafloxacin: Number of Treatment-emergent Adverse Events
Description: This study will evaluate the safety of the different regimens of finafloxacin. The safety outcome measures assessed are the following: vital signs, physical examinations, ECGs, haematology, biochemistry, urinalysis, adverse events and serious adverse events. Adverse events and serious adverse events will be documented throughout the study for each group (including comparator group and the incidence and severity of their occurrence will be compared between all groups. The results of all other safety outcome measures will be compared with the baseline values of each group to determine if significant changes occurred during the course of the study within one group. The results at the different visits will also be compared between the groups to identify significant differences between the 3 treatment groups.
Time Frame: Screening to Day 24
Population: Safety (SAF) population includes all subjects with at least one administration of study drug.
Measure: Number; unit: Treatment-emergent AEs
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days
Number analyzed (Participants) | 76 | 75 | 72
Treatment-emergent AEs | 70 | 51 | 70

6. Secondary Outcome: The Safety and Tolerability of Multiple Doses of Finafloxacin: Number of Participants Who Discontinued Due to TEAE
Description: as for outcome 5
Time Frame: Screening to day 24
Population: Safety (SAF) population includes all subjects with at least one administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days
Number analyzed (Participants) | 76 | 75 | 72
Participants | 7 | 2 | 4

ADVERSE EVENTS:
Time Frame: From screening to end-of-study visit, 24 - 28 days.
Arm/Group | Finafloxacin 5 Days | Finafloxacin 10 Days | Ciprofloxacin 10 Days
Serious Adverse Events (participants affected / at risk) | 3/76 | 4/75 | 1/72
Other Adverse Events (participants affected / at risk) | 29/76 | 19/75 | 29/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finafloxacin 5 Days (N=76) | Finafloxacin 10 Days (N=75) | Ciprofloxacin 10 Days (N=72)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Ovarian mucinous cystadenoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finafloxacin 5 Days (N=76) | Finafloxacin 10 Days (N=75) | Ciprofloxacin 10 Days (N=72)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 3 (5) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 4 (5) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (7) | 3 (3) | 6 (9)
Insomnia (Psychiatric disorders) | 3 (4) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Vomitting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Injection site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No